CLINICAL TRIAL: NCT01938300
Title: Magnesium and Rotational Thromboelastometry (ROTEM) in Colorectal Cancer Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Dr., Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Mg-ROTEM-colorectal ca
Record Dates: First submitted 2013-08-30; First posted 2013-09-10 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Magnesium (Experimental): Magnesium sulfate infusion during a operation period.
  Infusion regimen:
  1. Bolus 50 mg/kg of magnesium sulfate in 100 ml normal saline over 15 minutes
  2. Infusion 15 mg/kg/h of magnesium sulfate throughout the operation
  Interventions: Drug: Magnesium Sulfate
- Control (Placebo Comparator): administration of normal saline as a same volume of magnesium sulphate as a same method.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Magnesium Sulfate
  Arms: Magnesium
Drug: Normal saline
  Arms: Control

SUMMARY:
Magnesium sulphate is given to the patients during the colorectal cancer surgery under the hypothesis that it would attenuate the postoperative hypercoagulability. The investigators intend to characterize the changes of coagulation in colorectal cancer patients by using the point-of-care device after the infusion of magnesium sulphate.

ELIGIBILITY:
Inclusion Criteria:

* The patients undergoing a laparoscopic colorectal cancer surgery

Exclusion Criteria:

* Renal disease
* Hepatic disease
* Neuromuscular disease
* Coagulation disorder
* Cardiopulmonary disease

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change of maximum clot firmness (MCF) of FIBTEM | 1 day before a operation, 1 hour after finishing a operation, and a postopearative 3 day
Change of Clotting time (CT) of INTEM | 1 day before a operation, 1 hour after finishing a operation, and a postopearative 3 day
Change of Clot firmness time (CFT) of INTEM | 1 day before a operation, 1 hour after finishing a operation, and a postopearative 3 day
Change of Alpha angle of INTEM | 1 day before a operation, 1 hour after finishing a operation, and a postopearative 3 day
Change of MCF of INTEM | 1 day before a operation, 1 hour after finishing a operation, and a postopearative 3 day
Change of CT of EXTEM | 1 day before a operation, 1 hour after finishing a operation, and a postopearative 3 day
Change of CFT of EXTEM | 1 day before a operation, 1 hour after finishing a operation, and a postopearative 3 day
Change of Alpha angle of EXTEM | 1 day before a operation, 1 hour after finishing a operation, and a postopearative 3 day
Change of MCF of EXTEM | 1 day before a operation, 1 hour after finishing a operation, and a postopearative 3 day

SECONDARY OUTCOMES:
Change of Hemoglobin | 1 day before a operation, 1 hour after finishing a operation, and a postopearative 3 day
Change of Platelet count | 1 day before a operation, 1 hour after finishing a operation, and a postopearative 3 day
Change of International normalized ratio of prothrombin time | 1 day before a operation, 1 hour after finishing a operation, and a postopearative 3 day
Change of Activated partial thrombin time | 1 day before a operation, 1 hour after finishing a operation, and a postopearative 3 day
Change of Fibrinogen | 1 day before a operation, 1 hour after finishing a operation, and a postopearative 3 day

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea